CLINICAL TRIAL: NCT00153790
Title: The Effect of Soy Lecithin-derived N-oleoyl-phosphatidyl-ethanolamine (NOPE) and Green Tea-derived Epigallocatechin Gallate (EGCG) on Indices of Weight Loss and Appetite Suppression
Brief Title: LEAN Project: Weight Loss and Appetite Suppression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cooper Institute (Other)
Collaborators: Chemi Nutra (Unknown)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CI0151
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Weight Loss
Keywords: green tea; weight; women
MeSH Terms: conditions — Weight Loss; Body Weight

INTERVENTIONS:
Drug: PhosphoLean

SUMMARY:
The primary aim is to examine whether the intake of PhosphoLEAN is effective in aiding a cohort of women in losing weight. Participants taking the supplement will have significantly greater improvement in study outcomes than those taking the placebo.

DETAILED DESCRIPTION:
Participants will be randomized to either a control or treatment group taking the dietary supplement containing a soy lecithin-derived N-oleoyl-phosphatidyl-ethanolamine (NOPE) and caffeine free Green Tea-derived epigallocathchin gallate (EGCG) whose trade name is PhosphoLean. The outcome is to determine the effects on indices of weight loss and appetite suppression. Participants will return at 6, 12, and 16 weeks for clinical measures.

ELIGIBILITY:
Inclusion Criteria:

* 30-45 years, women, overweight or obese class I, premenopausal, maintain current diet and exercise regimen

Exclusion Criteria:

* pregnant or planning to become pregnant, currently have or history of cancer, heart disease, anemia, diabetes, depression

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2005-04; Study Completion 2006-05

PRIMARY OUTCOMES:
Weight Loss
Appetite Suppression

CONTACTS AND LOCATIONS:
Overall Officials: Conrad Earnest, PhD, Principal Investigator — The Cooper Institute
Locations (1):
- The Cooper Institute, Dallas, Texas, United States